CLINICAL TRIAL: NCT02780232
Title: A Randomized Controlled Trial of an Internet-based Program for Prevention and Early Intervention of Adolescent Depression
Brief Title: An Internet-based Program for Prevention and Early Intervention of Adolescent Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CES University (Other)
Collaborators: Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government); Universidad de Antioquia (Other); MIDAP Millennium Institute for Research in Depression and Personality (Unknown)
Responsible Party: Principal Investigator, Henry Daniel Espinosa Duque, MA, CES University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CES577
Record Dates: First submitted 2016-05-18; First posted 2016-05-23 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Depression
Keywords: Depression; Adolescence; Prevention; Early intervention; E-Mental Health
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based program (Experimental): Adolescents in the intervention will receive a tailored online program during 3 months.
  Adolescents interact with the program via a monitoring e-mail that they receive every two weeks (Monitoring) and a website which allows them to access a number of links.
  Interventions: Behavioral: Cuida tu animo / Care for your mood
- Treatment as usual (No Intervention): -Waiting list control group.

INTERVENTIONS:
Behavioral: Cuida tu animo / Care for your mood — CUIDA TU ÁNIMO is an online program to adolescents that provides information, education and support related to the care of the mood.
  Adolescents interact with the program via a monitoring e-mail that they receive every two weeks (Monitoring) and a website which allows them to access a number of links. The website have the following modules:
  1. What is 'CUIDA TU ÁNIMO': Description and definition of the program
  2. Psycho-educational information: Information about depression, its treatment, and opportunities for prevention
  3. How is your mood? (Monitoring): a) Online assessment of symptoms every two weeks during three months with the PHQ-3. b) Feedback
  4. Forums.
  5. Blog.
  6. Appointment (Chat or Phone call).
  7. Contact.
  Arms: Internet-based program

SUMMARY:
Major depression is a highly prevalent and severe mental disease. Interventions based on information and communication technologies (ICTs) generate innovative opportunities to prevent and to intervene early the depression in adolescents. In Colombia, there are few preventive mental health interventions scientifically oriented and seeking to demonstrate efficacy in context.

The purpose of this study is to determine whether an internet-based program is effective to prevent and to intervene early the depression in adolescents between 13 and 19 years of age in 8 schools of the Antioquia Region, Colombia .

Study design: A cluster-randomized clinical trial will be carried out with 600 adolescents. The efficacy, adherence, and acceptability of the internet-based program will be evaluated. A single-blind randomized controlled trial will be conducted with two arms, the intervention arm (n=300), which will receive an internet-based program for depression, and the TAU (Treatment As Usual) arm (n=300).

DETAILED DESCRIPTION:
Major depression is a highly prevalent and severe mental disease that negatively alters the lives of people, their families, and their social environment.

Organizations that promote mental health policies have recognized the potential of new information technologies for the prevention and treatment of mental disorders. In this direction, information and communication technologies (ICTs) generate opportunities for increasing patient well-being through the use of on-line software. Such programs often include interactivity, self-monitoring, information materials (sometimes in multimedia format), and exercises on problem solving, recognition and challenging of dysfunctional thoughts, scheduling of activities, behavioral experiments, and other psycho-educational activities.

In Colombia, there are few preventive mental health interventions scientifically oriented and seeking to demonstrate efficacy in context.

The purpose of this study is to determine whether an internet-based program is effective to prevent and to intervene early the depression in adolescents between 13 and 19 years of age in 8 schools in the Antioquia Region, Colombia.

Study design: A cluster-randomized clinical trial will be carried out with 600 adolescents. The efficacy, adherence, and acceptability of the internet-based program will be evaluated. A single-blind randomized controlled trial will be conducted with two arms, the intervention arm (n=300), which will receive an internet-based program for depression, and the TAU arm (n=300).

Follow-up times: T = 0 baseline, T= 3 months (post-intervention), T=12 months.

ELIGIBILITY:
Inclusion Criteria:

* Young students in schools of Antioquia between 6 and 11 high school degree, with internet access and available psychological service, foreseeing that moderate or severe depressive symptoms may be found.

Exclusion Criteria:

* Young students with high suicide risk defined by: score equal to or greater than 2 in question 9 of PHQ-9; students who are receiving at the time treatment with antidepressant drugs and / or currently attending psychotherapy.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-05-11 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Depressive Symptomatology at 3 months and 12 months | Baseline, 3 months, 12 months
  Depressive symptomatology measured with the Patient Health Questionnaire PHQ -9 [6]

SECONDARY OUTCOMES:
Change from Baseline in Health Related Quality of Life at 3 and 12 months | Baseline, 3 months, 12 months
  Health Related Quality of Life Questionnaire for Children and Young People KIDSCREEN-27 [7]
Change from Baseline in anxious symptoms at 3 and 12 months | Baseline, 3 months, 12 months
  Generalised Anxiety Disorder Assessment (GAD-7) [8]
Change from Baseline in of depression at 3 and 12 months | Baseline, 3 months, 12 months
  Self-Stigma of Depression Scale (SSDS) [9]

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Espinosa, MA, Principal Investigator — CES University
Locations (3):
- Colombia (3):
  - Institucion Educativa Villaflora, Medellín, Antioquia
  - Institucion Educativa El Pedregal, Medellín, Antioquia
  - Institución Educativa El Corazon, Medellín, Antioquia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sobocki P, Jonsson B, Angst J, Rehnberg C. Cost of depression in Europe. J Ment Health Policy Econ. 2006 Jun;9(2):87-98. PMID 17007486
- [Background] Vargas-Zea N, Castro H, Rodriguez-Paez F, Tellez D, Salazar-Arias R. Colombian Health System on its Way to Improve Allocation Efficiency-Transition from a Health Sector Reform to the Settlement of an HTA Agency. Value Health Reg Issues. 2012 Dec;1(2):218-222. doi: 10.1016/j.vhri.2012.09.004. Epub 2012 Dec 12. PMID 29702903
- [Background] Barney LJ, Griffiths KM, Christensen H, Jorm AF. The Self-Stigma of Depression Scale (SSDS): development and psychometric evaluation of a new instrument. Int J Methods Psychiatr Res. 2010 Dec;19(4):243-54. doi: 10.1002/mpr.325. PMID 20683846
- [Background] Fernández, J. & Gómez-Restrepo, C. Telepsiquiatría: innovación de la atención en salud mental. Una perspectiva general. Rev. Colomb. Psiquiat., 40 (3), 2011.
- [Background] Collins PY, Patel V, Joestl SS, March D, Insel TR, Daar AS; Scientific Advisory Board and the Executive Committee of the Grand Challenges on Global Mental Health; Anderson W, Dhansay MA, Phillips A, Shurin S, Walport M, Ewart W, Savill SJ, Bordin IA, Costello EJ, Durkin M, Fairburn C, Glass RI, Hall W, Huang Y, Hyman SE, Jamison K, Kaaya S, Kapur S, Kleinman A, Ogunniyi A, Otero-Ojeda A, Poo MM, Ravindranath V, Sahakian BJ, Saxena S, Singer PA, Stein DJ. Grand challenges in global mental health. Nature. 2011 Jul 6;475(7354):27-30. doi: 10.1038/475027a. No abstract available. PMID 21734685
- [Background] Lowe B, Decker O, Muller S, Brahler E, Schellberg D, Herzog W, Herzberg PY. Validation and standardization of the Generalized Anxiety Disorder Screener (GAD-7) in the general population. Med Care. 2008 Mar;46(3):266-74. doi: 10.1097/MLR.0b013e318160d093. PMID 18388841
- [Background] Moras, K. Twenty-five years of psychological treatment research on unipolar depression in adult outpatients: Introduction to the special section. Psychotherapy Research , 16 (5), 519-525, 2006.
- [Background] Proudfoot JG. Computer-based treatment for anxiety and depression: is it feasible? Is it effective? Neurosci Biobehav Rev. 2004 May;28(3):353-63. doi: 10.1016/j.neubiorev.2004.03.008. PMID 15225977
- [Background] Richardson LP, McCauley E, Grossman DC, McCarty CA, Richards J, Russo JE, Rockhill C, Katon W. Evaluation of the Patient Health Questionnaire-9 Item for detecting major depression among adolescents. Pediatrics. 2010 Dec;126(6):1117-23. doi: 10.1542/peds.2010-0852. Epub 2010 Nov 1. PMID 21041282
- [Background] KIDSCREEN Group Europe. The KIDSCREEN questionnaires. Quality of life questionnaires for children and adolescents- Handbook. Lengerich, Germany: Papst Science Publisher. 2006.